CLINICAL TRIAL: NCT02102347
Title: Effect of Phototherapy Incorporated Into an Exercise Program on Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Mcs, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24568013.0.0000.5511
Record Dates: First submitted 2014-03-29; First posted 2014-04-02 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Osteoarthritis of the Knee
Keywords: Physical Therapy Modalities; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Exercise; Phototherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- exercise group (Experimental): An exercise program will be performed to increase range of motion, improve motor learning and strengthen the muscles of the lower limb. The program will include exercises 2 times a week for four weeks. The first week the exercises will be performed with 2 sets of 15 repetitions and the remaining weeks 3 sets of 15 repetitions for each exercise. To exercise will be performed with the resistance of cinnamon, It will be recommended weight by 70% of one repetition maximum painless assigned individually per patient.
  Interventions: Other: exercise
- phototherapy group (Experimental): And, Phototherapy will be administered with a portable nine-diode cluster. The portable nine-diode cluster will be used overlapping three quadrants of the knee in random sequence: medial quadrant, lateral quadrant and posterior quadrant.with one 905-nm diode (mean power: 1 milliwatt ; peak power: 10 megawatt; spot size: 0.44 cm2), four 875-nm diodes (mean power of each diode: 17.5 milliwatt; spot size: 1 cm2) and four 670-nm diodes (mean power of each diode: 15 mW; spot size: 1 cm2); frequency: 1000 Hz; 300-second irradiation time in each quadrant; total energy: 39.3 Joules per quadrant. Phototherapy will be included in the exercises group.
  Interventions: Other: exercise; Other: Phototherapy
- Phototherapy placebo (Placebo Comparator): Phototherapy will be administered with a portable nine-diode cluster. The portable nine-diode cluster will be used overlapping three quadrants of the knee in random sequence: medial quadrant, lateral quadrant and posterior quadrant), with one 905-nm diode (mean power: 0 milliwatt; peak power: 0 watt; spot size: 0.44 cm2), four 875-nm diodes (mean power of each diode: 0 milliwatt; spot size: 1 cm2) and four 670-nm diodes (mean power of each diode: 0 milliwatt; spot size: 1 cm2); frequency: 0 Hz; 300-second irradiation time in each quadrant; total energy: 0 Joules per quadrant. Phototherapy will be included in the exercises group.
  Interventions: Other: exercise; Other: Phototherapy

INTERVENTIONS:
Other: exercise
Other: Phototherapy
  Arms: Phototherapy placebo; phototherapy group

SUMMARY:
The aim of the proposed study is to analyze the effect of the incorporation of phototherapy into a therapeutic exercise program on pain, functional capacity, range of motion, muscle strength in individuals with osteoarthritis of the knees. The participants will be allocated to different groups through a randomization process using opaque envelopes containing cards stipulating one of the three following groups: Group A (exercise protocol); Group B (exercise protocol + phototherapy protocol); and Group C (exercise protocol + placebo phototherapy protocol). Phototherapy will be performed on the knees diagnosed with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis of the knee (unilateral) according to criteria of the American College of Rheumatology
* age between 40 and 80 years
* either gender
* knee pain and functional disability for at least six months confirmed by historical medical.

Exclusion Criteria:

* Dementia
* neurological disorder (sensory or motor)
* cancer
* diabetes
* acute adverse health condition
* symptoms of osteoarthritis of the hip
* cardiopulmonary disease that impedes walking
* need for wheelchair or gait-assistance device
* and having received steroids through intra-articular injection or orally in the previous six months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
physical function | 9 months
  Using the Western Ontario and McMaster Universities Arthritis Index

SECONDARY OUTCOMES:
Maximum voluntary isometric contraction | 9 months
  A portable dynamometer will be used to assess muscle contraction.

OTHER OUTCOMES:
lower limb functionality | 9 months
  Using Extremity Functional Scale
pain | 9 months
  Numeric pain rating scale
level of pressure pain | 9 months
  threshold digital algometer
Timed up-and-go test | 9 months
  dynamic equilibrium
trunk stability | 9 months
  Functional reach test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Coelho Cde F, Leal-Junior EC, Biasotto-Gonzalez DA, Bley AS, de Carvalho Pde T, Politti F, Gonzalez Tde O, de Oliveira AR, Frigero M, Garcia MB, Dibai-Filho AV, Gomes CA. Effectiveness of phototherapy incorporated into an exercise program for osteoarthritis of the knee: study protocol for a randomized controlled trial. Trials. 2014 Jun 11;15:221. doi: 10.1186/1745-6215-15-221. PMID 24919587
- See also: Related Info — http://www.uninove.br